CLINICAL TRIAL: NCT01101126
Title: Disease Management Program for Chronic Obstructive Pulmonary Diseases in Maccabi Health Services
Brief Title: Disease Management in Asthma or Chronic Obstructive Pulmonary Disease (COPD) Patients
Acronym: ACDM-Maccabi
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: An excess of all-cause acute health services utilization in the intervention arm
Sponsor: Sheba Medical Center (Other Government)
Collaborators: Maccabi Healthcare Services, Israel (Other)
Responsible Party: Principal Investigator, Ofra Kalter-Leibovici MD, Dr., Sheba Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SHEBA-10-7741-OK-CTIL
Record Dates: First submitted 2010-04-08; First posted 2010-04-09 (Estimated); Last update posted 2015-01-21 (Estimated); Status verified 2015-01

CONDITIONS: Chronic Obstructive Pulmonary Disease (COPD); Asthma
Keywords: Chronic obstructive pulmonary disease (COPD); Asthma
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Asthma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Disease Management (Experimental): Comprehensive care delivered by designated nurses and pulmonologists, in collaboration with the primary practitioners and other healthcare professionals in the community
  Interventions: Other: Pulmonary disease management
- Unual care (Active Comparator): Care delivered by the primary practitioner with the advice of a consultant pulmonologist
  Interventions: Other: Usual care

INTERVENTIONS:
Other: Pulmonary disease management — Comprehensive pulmonary care including patient education of self-care, coordination of care, monitoring of patient adherence, providing advice in acute exacerbations
  Arms: Disease Management
Other: Usual care — Pulmonary disease is managed by the primary practitioner and a consultant pulmonologist
  Arms: Unual care

SUMMARY:
The purpose of this study is to determine whether disease management program is effective in preventing acute exacerbations in patients with unstable chronic obstructive pulmonary disease (COPD) or asthma.

DETAILED DESCRIPTION:
The aim of the present study is to test the efficacy of a comprehensive community disease management program in patients with unstable chronic obstructive pulmonary disease (COPD) or asthma. The intervention is delivered by designated nurses and pulmonologists, in collaboration with the primary practitioners and other healthcare professionals at the community, in the Jerusalem and the Lowland District of Maccabi Health Services in Israel.

The main purpose is to evaluate the effect of the intervention on the use acute care and emergency health services for acute exacerbation of the lung disease.

Secondary objectives include the evaluation of the effect of the intervention on quality of life, physical function, pulmonary function test, depression and all-cause mortality.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women
2. 40 years or older
3. Having unstable COPD or Asthma

Exclusion Criteria:

1. Significant LV dysfunction
2. Other severe chronic morbidity compromising short-term survival
3. Significant cognitive impairment or psychiatric disease
4. Bedridden
5. Homeless or no telephone connection

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 492 (Actual)
Dates: Start 2010-03; Primary Completion 2013-03 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Healthcare services utilization for acute exacerbations of pulmonary disease | Every 6 months during 1-3 years' follow-up
  The proportion of patients who, due to exacerbation of their COPD or asthma, have at least one out of hours visit to a "off-hour non-hospital based acute-care facilities", or a visit to a hospital emergency room, or a hospitalization within the two years of follow-up.

SECONDARY OUTCOMES:
Quality of life | Every 6 months during 1-3 years' follow-up
  Health-related quality of life
Pulmonary function tests | Every 6 months during 1-3 years' follow-up
  Pulmonary function tests
Physical function | Every 6 months during 1-3 years' follow-up
  6-minutes walk test assessment
Depression | Every 6 months during 1-3 years' follow-up
  PHQ-9 Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Meir Raz, M.D., Principal Investigator — Maccabi Healthcare Services, Israel; Ofra Kalter - Leibovici, M.D., Study Director — Sheba Medical Center
Locations (2):
- Israel (2):
  - Maccabi Pulmonary Clinic, Bat Yam
  - Maccabi Pulmonary Clinic, Holon